CLINICAL TRIAL: NCT06125483
Title: A Clinical Study of Low-dose Total Body Irradiation and Fludarabine/Busulfan/Melphalan as a Conditioning Regimen for Secondary Umbilical Cord Blood Transplantation in Patients With Hematological Malignancies Who Relapsed After Allo-HSCT
Brief Title: TBI/Flu/Bu/Mel Combined With Secondary UCBT in Patients With Hematological Malignancies Who Relapsed After Allo-HSCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOOCHOW-WXJ-2023-300
Record Dates: First submitted 2023-11-06; First posted 2023-11-09 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-09

CONDITIONS: Hematopoietic Malignancy; Relapse/Recurrence; Hematopoietic Stem Cell Transplantation
Keywords: Umbilical Cord Blood Transplantation; Conditioning Regimen; Secondary transplantation; Post-transplant Relapse
MeSH Terms: conditions — Hematologic Neoplasms; Recurrence | interventions — Cord Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 38 patients with hematological malignancies who received TBI/Flu/Bu/Mel combined with secondary UCBT (Experimental): Treatment stage : ( 1 ) conditioning : -7d, total body irradiation (TBI), 4Gy, 2 times ; -7d, semustine ( MECCNU ) 250mg / m2 ; -6d ~ -3d ; fludarabine ( Flu ) 30mg / m2 / d, ivgtt ; -6d ~ -5d, busulfan ( Bu ) 2.4mg / kg / d, 3 times a day, ivgtt ; -4d ~ -3d, melphalan ( Mel ) 40mg / m2 / d, ivgtt. ( 2 ) Transplantation : On day 0, unrelated umbilical cord blood ( TNC ≥ 2.3 × 107 / kg or CD34 + ≥ 1 × 105 / kg ) was transplanted, and the donor-recipient HLA matching degree was ≥ 6 / 10.
  Interventions: Procedure: Umbilical Cord Blood Transplantation

INTERVENTIONS:
Procedure: Umbilical Cord Blood Transplantation — Compared with peripheral blood stem cell transplantation (PBST), UCBT has a higher transplantation rate, as cord blood stem cells are more primitive. Since the first successful umbilical cord blood transplantation (UCBT) in a child with severe Fanconi anemia reported by Gluckman et al. in France in 1988, cord blood has been widely used as a graft source of hematopoietic stem cells for the treatment of hematological diseases. The first sibling UCBT for leukemia was performed successfully by Professor Yongping Song in China, who played a pioneering role in the development of UCBT for leukemia in China. On the basis of previous research, TBI/Flu/Bu/Mel combined with UCBT is safe and feasible for the treatment of patients with malignant hematological diseases who experienced post-transplant relapse, which has enormous potential to improve patient outcomes.
  Other Names: Total Body Irradiation/Fludarabine/Busulfan/Melphalan

SUMMARY:
About 33% of patients with myeloid or lymphoid malignancies experience relapse with HLA loss after haplo-HSCT. Due to the specificity of HLA-loss relapse, the 2019 European Society for Blood and Marrow Transplantation (EBMT) pointed out that for diagnosed HLA-loss patients, it is recommended to use different HLA-haploidentical donors, and lymphocyte infusions from the original donor cannot improve the prognosis. Clinical studies have found that second transplantation can achieve prolonged disease-free survival than chemotherapy for patients with HLA loss, and it may be an effective treatment strategy for these patients.

However, due to the high standard of second hematopoietic stem cell transplantation (HSCT), not all patients can find suitable donors. Since the first successful application of umbilical cord blood transplantation (UCBT) by Gluckman et al. in France in 1988 for the treatment of Fanconi anemia, umbilical cord blood (UCB) has been widely used as a reliable source for HSCT in the treatment of hematological diseases. In 1998, Professor Yongping Song led the first successful UCBT in the treatment of leukemia, opening up the path of it in China. Compared with peripheral blood stem cell transplantation (PBST), UCBT has a higher engraftment rate. UCB contains more primitive and purer stem cells than bone marrow hematopoietic stem cells. UCBT can be performed with only 4 HLA matches, and the degree of rejection, the risk of disease relapse, and the incidence of chronic graft-versus-host disease (cGVHD) are all relatively low, greatly improving the survival of patients.

Although UCBT has been a potential treatment for second transplantation, the effective conditioning regimen is still under discussion. Improving the incidence of engraftment , the tolerance of conditioning, and reducing transplant-related mortality (TRM) are issues of great concern in second transplantation. A standard RIC regimen composed of fludarabine (200mg/m2) combined with cyclophosphamide (50mg/kg) and 2Gy or 3Gy total body irradiation (TBI) is the most common conditioning regimen used in UCBT. Although the tolerance of this RIC is acceptable, the relapse rate after transplantation is relatively high, and the implantation failure rate is also high in high-risk populations. The inclusion of thiotepa (10mg/kg) combined with fludarabine, cyclophosphamide, and 4Gy TBI in an intensified version of the RIC regimen has improved the engraftment rate without increasing TRM. In addition, studies have also confirmed that increasing the dose of TBI can improve engraftment in transplant recipients at high risk of UCBT failure. The fludarabine/busulfan/melphalan (Flu/Bu/Mel) conditioning regimen was first used for salvaging UCBT in unresponsive hematological malignancies in 2016 and achieved good clinical outcomes. Subsequently, several transplant centers in Japan adopted the Flu/Bu/Mel conditioning regimen for UCBT and confirmed that, compared with the Flu/Bu4 regimen, it not only improved overall survival (OS) but also reduced disease relapse rate without increasing TRM. A recent multicenter retrospective study of UCBT in patients with acute myeloid leukemia in remission found that compared with the TBI/Cy conditioning regimen, the Flu/Bu/Mel conditioning regimen improved the engraftment rate and exerted the GVL effect, reducing NRM and improving OS.

Based on the above, TBI/Flu/Bu/Mel as a conditioning regimen for secondary UCBT in patients with hematological malignancies who relapsed after allo-HSCT is safe and feasible, and is expected to improve the prognosis of these patients. Therefore, based on existing clinical experience with research evidence, our center plans to conduct a clinical study of low-dose TBI and FBM as a conditioning regimen for secondary UCBT in patients with hematological malignancies who relapsed after allo-HSCT, observing the improvement in the cumulative incidence of engraftment, disease relapse, GVHD, and survival rate in patients who received this regimen.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is an effective treatment for hematological malignancies, and post-transplant relapse is the primary cause of death. The optimal treatment strategy for leukemia relapse after allo-HSCT is still unclear, and the treatment options for these relapsed patients are limited. They mainly include chemotherapy, targeted therapy, donor lymphocyte infusion, immune checkpoint inhibitors, chimeric antigen receptor T-cell therapy (CAR-T), bispecific antibodies, and secondary hematopoietic stem cell transplantation. Although many factors may contribute to post-transplant relapse, such as insensitivity of leukemia cells to the conditioning regimen, in most cases, the leukemia cells escape immune surveillance by donor T cells, leading to 'immune escape'. The source of T cells is one of the main driving factors for the graft-versus-leukemia (GVL) effect after allo-HSCT. Therefore, all the typical mechanisms of immune escape and tumor immunity in relapse after allo-HSCT will ultimately eliminate the interaction between T cells and tumors. This may be due to the mechanisms of patient-specific HLA loss in dual relapse: cytotoxic T lymphocytes (CTL) reduce the GVL effect of allogeneic immunity through non-MHC-restricted HLA; important HLA locus loss reduces leukemia antigen presentation and cannot induce CTL production, directly leading to immune escape.

In traditional relapsed patients, only 10-32% of acute myeloid leukemia (AML) patients can achieve remission again through treatment, and the prognosis is worse in acute lymphocytic leukemia (ALL) patients, with a median survival of about 10 months. Yaara Yerushalmi et al. conducted a retrospective analysis of 407 patients with post-transplant relapse, among which 62 patients underwent secondary HSCT. The 5-year overall survival (OS) rate in the secondary transplantation group reached 25%, while it was only 7% in the non-secondary transplantation group of 345 patients. Secondary HSCT improves the prognosis of these patients.

UCB contains abundant hematopoietic stem cells, endothelial progenitor cells, mesenchymal stem cells, and other types of stem/progenitor cells, as well as immune cells such as natural killer cells and Treg cells. These stem/progenitor cells have strong self-renewal and proliferation ability, low immunogenicity, and could secrete various hematopoietic growth factors that act on myeloid cells, granulocytes, etc., facilitating hematopoietic reconstruction and recovery. They include platelet growth factor, erythropoietin, stem cell factor, and various interleukins. The content of various cytokines such as stem cell factor, IL-6, and IL-11 in UCB is much higher than that in peripheral blood. The potential mechanism of UCB in hematological disease treatment is largely the result of the interaction between various growth factors and stem/progenitor cells and the body.

The team led by Professor Sun Zimin at the Anhui Provincial Hospital was the first to use UCBT to treat patients with AML. They found that the incidence of cGVHD and relapse in patients significantly decreased, while the survival rate of patients without GVHD or relapse significantly improved, greatly improving the OS of patients. UCBT has also been widely applied in other malignant diseases such as ALL, malignant lymphoma, and multiple myeloma (MM). In 2017, an adult AML patient was successfully treated with UCBT at Wuhan Central Hospital and discharged to resume normal life. In 2020, a 14-year-old patient with myeloproliferative neoplasms was treated with UCBT at Tai'an Central Hospital. The patient had a mild rejection reaction after transplantation but achieved good recovery and was eventually safely discharged. Since April 2021, the Seventh Hospital of Zhongshan has successfully completed 10 cases of UCBT, including patients with high body weight (85kg), highly positive panel reactive antibodies (PRA), or second transplantation. The overall response rate is 100%, with the longest disease-free survival time being 2 years, only 1 case of severe GVHD, no TRM, or relapse. Therefore, UCBT has tremendous potential in the second HSCT.

The conditioning regimen is a key link in transplantation, and a reduced-intensity conditioning (RIC) regimen has improved the second transplantation tolerance in patients due to its relatively low toxicity. Whether after autologous transplantation or allo-HSCT, a reduced-intensity conditioning regimen has been proven in multiple studies to reduce non-relapse mortality and relapse rate in second transplantation (RIC2 HSCT). A retrospective study which conducted by EBMT included 234 patients who underwent a RIC regimen for second transplantation, with a 2-year non-relapse mortality rate of 22.4% and a relapse rate of 63.9%.

ELIGIBILITY:
Inclusion Criteria:

1. Gender is not limited, patients between 10 to 65 years old (including critical value);
2. According to the WHO diagnostic criteria, the diagnosis of hematological malignancies ( acute lymphoblastic leukemia, acute / chronic myeloid leukemia, etc. ) was confirmed by bone marrow puncture or biopsy after allogeneic hematopoietic stem cell transplantation. The definition of relapse includes the proportion of bone marrow blast cells > 5 %, blast cells in peripheral blood ( excluding the use of G-CSF and GM-CSF ), or extramedullary leukemia infiltration;
3. Planned to received umbilical cord blood transplantation;
4. The indexes of cardiac function, liver and kidney function were within the following limits:(1) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3× Upper limit of normal (ULN); (2)Total bilirubin ≤ 3×ULN; (3) Serum creatinine ≤ 2×ULN or creatinine clearance ≥ 40mL/min; (4) Left ventricular ejection fraction (LVEF) as measured by echocardiography or multi-gated acquisition (MUGA) scan is within the normal range (> 50%);
5. Umbilical cord blood with HLA match ≥ 6/10;
6. Expected survival ≥3 months;
7. Karnofsky (KPS) score ≥60%, Eastern Tumor Cooperative group (ECOG) status ≤ 2;
8. Patient fully understood the nature of the study, and voluntarily participates and signs informed consent.

Exclusion Criteria:

1. Patients had serious adverse reactions to investigational drugs such as allergies;
2. Patient was complicated with pulmonary infection, which was confirmed by imaging to be progressive;
3. Patients with hypertension, ventricular arrhythmia requiring clinical intervention, acute coronary syndrome, congestive heart failure, stroke, or other grade III or higher cardiovascular events within 6 months;
4. Patients with active viral infections, including HIV, HBV, HCV, TP;
5. Pregnant or lactating patients;
6. The patient is currently participating in another clinical studies;
7. Patients deemed unsuitable for inclusion by other investigators.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | within 1 year following UCBT
  We estimated OS from the time of transplant until the date of death of any cause or last follow-up for patients still alive.

SECONDARY OUTCOMES:
The cumulative incidence of engraftment | Neutrophil engraftment: on day 28±7 following UCBT; Platelet engraftment: on day 100±7 following UCBT
  Neutrophil and platelet engraftment is defined as the first occurrence of 3 consecutive days with an absolute neutrophil count of at least 0.5×109/L and a platelet count of over 20×109/L for 7 consecutive days without transfusion support.
The cumulative incidence and severity of pre-engraftment syndrome (PES) | on day 28±7 following UCBT
  Pre-engraftment syndrome (PES) is a condition occurring after umbilical cord blood transplantation (UCBT) characterized by fever and erythematous skin rash prior to neutrophil engraftment.
The cumulative incidence and grade of graft-versus-host disease (GVHD) | within 100 days following UCBT (acute GVHD); within 1 year following UCBT (chronic GVHD)
  Graft-versus-host disease (GVHD) is a medical complication following the receipt of transplanted tissue from a genetically different person.
The cumulative incidence of relapse | within 1 year following UCBT
  We defined relapse as any clinical evidence of progression or recurrence of original diseases.
The cumulative incidence of non-relapsed mortality (NRM) | within 1 year following UCBT
  Non-relapsed mortality was defined as mortality due to any cause other than disease progression or relapse.
The time of disease-free survival | within 1 year following UCBT
  Disease-free survival (DFS) is defined as the time from randomization to recurrence of tumor or death.
The cumulative incidence of adverse event | within 1 year following UCBT
  Following extraction of the tumor, a blood vessel burst causing increased blood loss during the procedure, an adverse event the surgeon did not expect.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojin Wu, Prof., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow university, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Cao XY, Zhang JP, Zhao YL, Xiong M, Zhou JR, Lu Y, Sun RJ, Wei ZJ, Liu DY, Zhang X, Yang JF, Lu P. Analysis benefits of a second Allo-HSCT after CAR-T cell therapy in patients with relapsed/refractory B-cell acute lymphoblastic leukemia who relapsed after transplant. Front Immunol. 2023 Jul 4;14:1191382. doi: 10.3389/fimmu.2023.1191382. eCollection 2023. PMID 37469510
- [Background] de Lima M, Porter DL, Battiwalla M, Bishop MR, Giralt SA, Hardy NM, Kroger N, Wayne AS, Schmid C. Proceedings from the National Cancer Institute's Second International Workshop on the Biology, Prevention, and Treatment of Relapse After Hematopoietic Stem Cell Transplantation: part III. Prevention and treatment of relapse after allogeneic transplantation. Biol Blood Marrow Transplant. 2014 Jan;20(1):4-13. doi: 10.1016/j.bbmt.2013.08.012. Epub 2013 Sep 7. PMID 24018392
- [Background] Christopeit M. When is second allogeneic HSCT for relapse of acute leukaemia an option? Bone Marrow Transplant. 2016 Feb;51(2):184-5. doi: 10.1038/bmt.2015.285. Epub 2015 Dec 7. No abstract available. PMID 26642335
- [Background] Rovatti PE, Gambacorta V, Lorentino F, Ciceri F, Vago L. Mechanisms of Leukemia Immune Evasion and Their Role in Relapse After Haploidentical Hematopoietic Cell Transplantation. Front Immunol. 2020 Feb 25;11:147. doi: 10.3389/fimmu.2020.00147. eCollection 2020. PMID 32158444
- [Background] Crucitti L, Crocchiolo R, Toffalori C, Mazzi B, Greco R, Signori A, Sizzano F, Chiesa L, Zino E, Lupo Stanghellini MT, Assanelli A, Carrabba MG, Marktel S, Marcatti M, Bordignon C, Corti C, Bernardi M, Peccatori J, Bonini C, Fleischhauer K, Ciceri F, Vago L. Incidence, risk factors and clinical outcome of leukemia relapses with loss of the mismatched HLA after partially incompatible hematopoietic stem cell transplantation. Leukemia. 2015 May;29(5):1143-52. doi: 10.1038/leu.2014.314. Epub 2014 Nov 5. PMID 25371177
- [Background] Arnold PY. Review: HLA loss and detection in the setting of relapse from HLA-mismatched hematopoietic cell transplant. Hum Immunol. 2022 Oct;83(10):712-720. doi: 10.1016/j.humimm.2022.03.001. Epub 2022 Mar 11. PMID 35287976
- [Background] Wu H, Shi J, Luo Y, Yu J, Lai X, Liu L, Fu H, Ouyang G, Xu X, Xiao H, Huang H, Zhao Y. Assessment of Patient-Specific Human Leukocyte Antigen Genomic Loss at Relapse After Antithymocyte Globulin-Based T-Cell-Replete Haploidentical Hematopoietic Stem Cell Transplant. JAMA Netw Open. 2022 Apr 1;5(4):e226114. doi: 10.1001/jamanetworkopen.2022.6114. PMID 35385089
- [Background] Mielcarek M, Storer BE, Flowers ME, Storb R, Sandmaier BM, Martin PJ. Outcomes among patients with recurrent high-risk hematologic malignancies after allogeneic hematopoietic cell transplantation. Biol Blood Marrow Transplant. 2007 Oct;13(10):1160-8. doi: 10.1016/j.bbmt.2007.06.007. Epub 2007 Aug 3. PMID 17889352
- [Background] Schmid C, Labopin M, Nagler A, Niederwieser D, Castagna L, Tabrizi R, Stadler M, Kuball J, Cornelissen J, Vorlicek J, Socie G, Falda M, Vindelov L, Ljungman P, Jackson G, Kroger N, Rank A, Polge E, Rocha V, Mohty M; Acute Leukaemia Working Party of the European Group for Blood and Marrow Transplantation (EBMT). Treatment, risk factors, and outcome of adults with relapsed AML after reduced intensity conditioning for allogeneic stem cell transplantation. Blood. 2012 Feb 9;119(6):1599-606. doi: 10.1182/blood-2011-08-375840. Epub 2011 Dec 13. PMID 22167752
- [Background] Yerushalmi Y, Shem-Tov N, Danylesko I, Canaani J, Avigdor A, Yerushalmi R, Nagler A, Shimoni A. Second hematopoietic stem cell transplantation as salvage therapy for relapsed acute myeloid leukemia/myelodysplastic syndromes after a first transplantation. Haematologica. 2023 Jul 1;108(7):1782-1792. doi: 10.3324/haematol.2022.281877. PMID 36475520
- [Background] Gluckman E, Broxmeyer HA, Auerbach AD, Friedman HS, Douglas GW, Devergie A, Esperou H, Thierry D, Socie G, Lehn P, et al. Hematopoietic reconstitution in a patient with Fanconi's anemia by means of umbilical-cord blood from an HLA-identical sibling. N Engl J Med. 1989 Oct 26;321(17):1174-8. doi: 10.1056/NEJM198910263211707. No abstract available. PMID 2571931
- [Background] Ehrhart J, Sanberg PR, Garbuzova-Davis S. Plasma derived from human umbilical cord blood: Potential cell-additive or cell-substitute therapeutic for neurodegenerative diseases. J Cell Mol Med. 2018 Dec;22(12):6157-6166. doi: 10.1111/jcmm.13898. Epub 2018 Oct 18. PMID 30334335
- [Background] Sun HP, Zhang X, Chen XH, Zhang C, Gao L, Feng YM, Peng XG, Gao L. Human umbilical cord blood-derived stromal cells are superior to human umbilical cord blood-derived mesenchymal stem cells in inducing myeloid lineage differentiation in vitro. Stem Cells Dev. 2012 Jun 10;21(9):1429-40. doi: 10.1089/scd.2011.0348. Epub 2011 Dec 5. PMID 22023173
- [Background] Sanchez-Petitto G, Rezvani K, Daher M, Rafei H, Kebriaei P, Shpall EJ, Olson A. Umbilical Cord Blood Transplantation: Connecting Its Origin to Its Future. Stem Cells Transl Med. 2023 Mar 3;12(2):55-71. doi: 10.1093/stcltm/szac086. PMID 36779789
- [Background] Zheng CC, Zhu XY, Tang BL, Zhang XH, Zhang L, Geng LQ, Liu HL, Sun ZM. Clinical separation of cGvHD and GvL and better GvHD-free/relapse-free survival (GRFS) after unrelated cord blood transplantation for AML. Bone Marrow Transplant. 2017 Jan;52(1):88-94. doi: 10.1038/bmt.2016.182. Epub 2016 Jul 4. PMID 27376453
- [Background] Foran JM, Pavletic SZ, Logan BR, Agovi-Johnson MA, Perez WS, Bolwell BJ, Bornhauser M, Bredeson CN, Cairo MS, Camitta BM, Copelan EA, Dehn J, Gale RP, George B, Gupta V, Hale GA, Lazarus HM, Litzow MR, Maharaj D, Marks DI, Martino R, Maziarz RT, Rowe JM, Rowlings PA, Savani BN, Savoie ML, Szer J, Waller EK, Wiernik PH, Weisdorf DJ. Unrelated donor allogeneic transplantation after failure of autologous transplantation for acute myelogenous leukemia: a study from the center for international blood and marrow transplantation research. Biol Blood Marrow Transplant. 2013 Jul;19(7):1102-8. doi: 10.1016/j.bbmt.2013.04.022. Epub 2013 Apr 28. PMID 23632091
- [Background] Shaw BE, Mufti GJ, Mackinnon S, Cavenagh JD, Pearce RM, Towlson KE, Apperley JF, Chakraverty R, Craddock CF, Kazmi MA, Littlewood TJ, Milligan DW, Pagliuca A, Thomson KJ, Marks DI, Russell NH. Outcome of second allogeneic transplants using reduced-intensity conditioning following relapse of haematological malignancy after an initial allogeneic transplant. Bone Marrow Transplant. 2008 Dec;42(12):783-9. doi: 10.1038/bmt.2008.255. Epub 2008 Aug 25. PMID 18724393
- [Background] Vrhovac R, Labopin M, Ciceri F, Finke J, Holler E, Tischer J, Lioure B, Gribben J, Kanz L, Blaise D, Dreger P, Held G, Arnold R, Nagler A, Mohty M; Acute Leukemia Working Party of the European Society for Blood and Marrow Transplantation (EBMT). Second reduced intensity conditioning allogeneic transplant as a rescue strategy for acute leukaemia patients who relapse after an initial RIC allogeneic transplantation: analysis of risk factors and treatment outcomes. Bone Marrow Transplant. 2016 Feb;51(2):186-93. doi: 10.1038/bmt.2015.221. Epub 2015 Oct 5. PMID 26437057
- [Background] Brunstein CG, Barker JN, Weisdorf DJ, DeFor TE, Miller JS, Blazar BR, McGlave PB, Wagner JE. Umbilical cord blood transplantation after nonmyeloablative conditioning: impact on transplantation outcomes in 110 adults with hematologic disease. Blood. 2007 Oct 15;110(8):3064-70. doi: 10.1182/blood-2007-04-067215. Epub 2007 Jun 14. PMID 17569820
- [Background] Sharma P, Pollyea DA, Smith CA, Purev E, Kamdar M, Haverkos B, Sherbenou D, Rabinovitch R, Hammes A, Gutman JA. Thiotepa-Based Intensified Reduced-Intensity Conditioning Adult Double-Unit Cord Blood Hematopoietic Stem Cell Transplantation Results in Decreased Relapse Rate and Improved Survival Compared with Transplantation Following Standard Reduced-Intensity Conditioning: A Retrospective Cohort Comparison. Biol Blood Marrow Transplant. 2018 Aug;24(8):1671-1677. doi: 10.1016/j.bbmt.2018.04.019. Epub 2018 Apr 21. PMID 29684565
- [Background] Ostronoff F, Milano F, Gooley T, Gutman JA, McSweeney P, Petersen FB, Sandmaier BM, Storb R, Delaney C. Double umbilical cord blood transplantation in patients with hematologic malignancies using a reduced-intensity preparative regimen without antithymocyte globulin. Bone Marrow Transplant. 2013 Jun;48(6):782-6. doi: 10.1038/bmt.2012.243. Epub 2012 Dec 17. PMID 23241738
- [Background] Yamamoto H, Uchida N, Yuasa M, Kageyama K, Ota H, Kaji D, Nishida A, Ishiwata K, Takagi S, Tsuji M, Asano-Mori Y, Yamamoto G, Izutsu K, Masuoka K, Wake A, Yoneyama A, Makino S, Taniguchi S. A Novel Reduced-Toxicity Myeloablative Conditioning Regimen Using Full-Dose Busulfan, Fludarabine, and Melphalan for Single Cord Blood Transplantation Provides Durable Engraftment and Remission in Nonremission Myeloid Malignancies. Biol Blood Marrow Transplant. 2016 Oct;22(10):1844-1850. doi: 10.1016/j.bbmt.2016.06.017. Epub 2016 Jun 21. PMID 27345142
- [Background] Shimomura Y, Hara M, Yamamoto H, Uchida N, Kawakita T, Ashida T, Takada S, Ikeda T, Morishige S, Maruyama Y, Wake A, Ichinohe T, Fukuda T, Takanashi M, Atsuta Y, Ishikawa T. Adding melphalan to fludarabine and a myeloablative dose of busulfan improved survival after allogeneic hematopoietic stem cell transplantation in a propensity score-matched cohort of hematological malignancies. Bone Marrow Transplant. 2021 Jul;56(7):1691-1699. doi: 10.1038/s41409-021-01217-w. Epub 2021 Mar 3. PMID 33658646
- [Background] Mizuno S, Takami A, Kawamura K, Shimomura Y, Arai Y, Konuma T, Ozawa Y, Sawa M, Ota S, Takahashi S, Anzai N, Hiramoto N, Onizuka M, Nakamae H, Tanaka M, Murata M, Kimura T, Kanda J, Fukuda T, Atsuta Y, Yanada M. Favorable Outcome with Conditioning Regimen of Flu/Bu4/Mel in Acute Myeloid Leukemia Patients in Remission Undergoing Cord Blood Transplantation. Transplant Cell Ther. 2022 Nov;28(11):775.e1-775.e9. doi: 10.1016/j.jtct.2022.07.026. Epub 2022 Aug 1. PMID 35921987